CLINICAL TRIAL: NCT02722655
Title: Characteristics and Evolution of Diabetes Mellitus in Mexican Children: Cohort Study
Brief Title: Cohort of Mexican Children With Diabetes Mellitus (CMC-DM)
Acronym: CMC-DM
Status: Recruiting | Type: Observational
Sponsor: Hospital Regional de Alta Especialidad del Bajio (Other)
Responsible Party: Principal Investigator, Maria Lola Evia-Viscarra, Pediatric Endocrinologist, Hospital Regional de Alta Especialidad del Bajio
Other Study IDs: 2015-018
Record Dates: First submitted 2016-03-18; First posted 2016-03-30 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Diabetes Mellitus
Keywords: Pediatrics
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Type 1 diabetes mellitus: Sudden onset of symptoms and non-overweight/obese
- Type 2 diabetes mellitus: Insidious onset of symptoms and overweight/obese
- Type 1.5 diabetes mellitus: Overlap of type 1 and type2 diabetes mellitus clinical characteristics
- Other types of diabetes mellitus: According American Diabetes Association criteria

SUMMARY:
The aim of this study is the identification of complications in diabetes mellitus pediatric patients and to compare the clinical, anthropometric, and biochemical characteristics between children in the different types of diabetes mellitus.

DETAILED DESCRIPTION:
Diabetes mellitus is characterized by hyperglycemia resulting from defects in insulin secretion and/or insulin resistance in target tissues. This study identify the influence of pathogenic factors on the evolution of diabetes mellitus and in the presence of chronic complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosis of diabetes mellitus

Exclusion Criteria:

-

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children and adolescents (boys and girls) from 1 months to 17 years of age that had recently been diagnosed with diabetes mellitus.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2008-03; Primary Completion 2020-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Diabetic retinopathy | year 3
  A microvascular complication determined by ophthalmological evaluation
Peripheral diabetic neuropathy | year 5
  A microvascular complication determined by neurological exam in either foot
Nerve damage | year 5
  A microvascular complication determined by nerve conduction study in either foot
Microalbuminuria | annual
  A microvascular complication determined by urine albumin excretion >= 30 mg/day
Cardiac function | year 5
  A cardiovascular risk indicator determined by echocardiogram
Cognitive evaluation | year 3
  Determined by scores on the Mini-Mental State Examination
Intelligence quotient evaluation | year 3
  Determined by Intelligence quotient test

SECONDARY OUTCOMES:
Body composition | annual
  Determined by body mass index (BMI) percentiles computed from physical measurements of height and weight and corresponding percentile tables
Glycemic control | annual
  Determined by HbA1c
Beta cell function | annual
  Determined by fasting C peptide
Pancreatic autoimmunity | onset of diabetes
  Determined by pancreas autoantibodies
Insulin resistance | annual
  Determined by insulin sensitivity
Alpha cell function | year 5
  Determined by glucagon
Hyperlipidemia | annual
  Determined by lipid profile
Hypothyroidism | annual
  Determined by thyroid profile
Hypertension | annual
  Determined by collection of systolic and diastolic blood pressure and calculation of their percentile values

CONTACTS AND LOCATIONS:
Overall Officials: María L Evia-Viscarra, Principal Investigator — Department of Pediatric Endocrinology, Hospital Regional de Alta Especialidad del Bajío
Locations (1):
- Hospital Regional de Alta Especialidad del Bajío, León, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Evia-Viscarra ML, Guardado-Mendoza R, Rodea-Montero ER. Clinical and Metabolic Characteristics among Mexican Children with Different Types of Diabetes Mellitus. PLoS One. 2016 Dec 16;11(12):e0168377. doi: 10.1371/journal.pone.0168377. eCollection 2016. PMID 27992493